CLINICAL TRIAL: NCT06257407
Title: Perioperative Hemostasis Management in Liver Transplantation
Acronym: HEMOTRANSPLANT
Status: Recruiting | Type: Observational
Sponsor: Société Française d'Anesthésie et de Réanimation (Other)
Collaborators: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Responsible Party: Sponsor
Other Study IDs: HEMOTRANSPLANT / 2022-12
Record Dates: First submitted 2024-01-31; First posted 2024-02-14 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Liver Transplant; Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults Patients with Liver transplant: No intervention during this observational study. Patient who meet the inclusion criteria will be included

SUMMARY:
Liver transplantation (LT) is a surgery with risk of bleeding. Several risk factors have been identified: complex dissection, portal hypertension, history of ascites fluid infections, history of surgical procedures, pre-existing complex hemostatic disorders and those acquired during the procedure. Diffuse bleeding can occur at any time during the 3 phases of surgery: dissection, anhepatic and neohepatic. However, intraoperative bleeding and transfusion requirements remain difficult to predict. Current predictive models are based in particular on preoperative characteristics and do not take into account the course and different phases of the operation.

The need for transfusions has largely decreased over the last 20 years, and currently around 20-25% of patients are transfused (transfusion of at least 1 blood product during LT). However, massive transfusion is necessary in 10% of LT. The European Society of Anaesthesiology (ESA) has issued recommendations on the management of severe bleeding during surgery. However, these recommendations are not specific to LT. Moreover, transfusion strategies vary widely from one center to another. The implementation of protocols within teams dedicated to LT has led to a reduction in bleeding and transfusion, with or without the use of viscoelastic testing.

Intraoperative bleeding and transfusion requirements, as well as postoperative thromboembolic complications, remain difficult to predict. Predictive models of bleeding risk have been developed, but they are based solely on preoperative characteristics and do not take into account the course and various phases of the operation. In addition, new methods such as Bayesian inference or machine learning have been developed, and seem capable of providing different information from that obtained by conventional models.

The overall aim of this prospective multicenter observational study is to investigate the risk factors for bleeding and thrombosis in per- and post-operative LT using different predictive methods, and to describe the management of bleeding and post-operative anticoagulation in metropolitan France.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or over
* Liver transplant patient

Exclusion Criteria:

* Multi-organ transplantation
* Protected populations: under guardianship or curatorship
* Patients not affiliated to a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver transplant patient
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Determine factors that predict the number of red blood cells packed (pRBCs) transfused intraoperatively in LT | number of pRBCs transfused during surgery
  Number of intraoperative pRBCs transfused

SECONDARY OUTCOMES:
Determine factors predicting transfusion of more than 2 pRBCs intraoperatively | During surgery
  (qualitative binary) transfusion of more than 2 intraoperative RBCs (Y/N)
Determine the predictive factors for intraoperative transfusion of RBCs for LT | During surgery
  (qualitative binary) intraoperative use of packed red blood cells (Y/N)
Determine the predictive factors of the number of RBCs transfused at each phase of LT | During surgery
  (quantitative) number of pRBCs transfused during each of the 3 phases of LT
Determine factors predicting intraoperative bleeding volume in LT | During surgery
  intraoperative bleeding volume
Determine haemoglobin mass loss in patients not receiving intraoperative pRBC transfusion of LT | During surgery
  Haemoglobin mass loss
Describe haemostatic tests (conventional biological and viscoelastic) carried out intraoperatively on LT. By listing all haemostatic tests performed | During surgery
  Haemostatic tests performed
Describe the use of blood products, blood-derived medicinal products and antifibrinolytics administered during each phase of LT and during the first 24 hours postoperatively. By listing all products administered. | During surgery
  Blood products, blood-derived medicinal products, antifibrinolytics
Determine the factors predicting the number of RBCs transfused within 24 hours post-LT | During 24 hours post-LT
  (quantitative) number of RBCs transfused in the 24 hours post-LT
To explore the links between bleeding or transfusion and the results of haemostatic tests (conventional biological and viscoelastic) in peri-operative LT. By comparing occurance of bleeding or transfusion and values of haemostatic tests. | During operation
  Results of haemostatic tests performed after bleeding or transfusion
Describe the post-operative use of anti-aggregants and anticoagulants drugs in LT | During the first 30 days postoperative LT
  Listing of Antiaggregation and thromboprophylaxis used
Describe postoperative venous thrombotic events (deep vein thrombosis, pulmonary embolism, portal thrombosis) and arterial (graft artery thrombosis) during the first 30 days postoperative LT | During the first 30 days postoperative LT
  Thrombotic complications
Measure the possible effect of the various pro- and antihaemostatic treatments on haemorrhagic and thrombotic complications in the first 30 days after LT surgery | During the first 30 days postoperative LT
  Thrombotic complications and haemorrhagic complications
Explore the links between thombothic events and the results of hemostatic tests (common biological tests and viscoelastic tests) | thombotic events observed during the first 30 days postoperative LT
  Results of hemostatic tests performed during thrombothic events

CONTACTS AND LOCATIONS:
Overall Officials: WEISS, MD, Principal Investigator — Hôpital Beaujon
Locations (16):
- France (16):
  - Chru Minjoz, Besançon
  - CHU Estaing, Clermont
  - Hôpital Beaujon, Clichy
  - CHU Grenoble Alpes, Grenoble
  - CHU Claude Huriez, Lille
  - Hôpital de la Croix-Rousse, Lyon
  - CHU La Timone, Marseille
  - Hôpital St Eloi, Montpellier
  - Hôpital De L'Archet 2, Nice
  - CHU Pitié-Salpêtrière, Paris
  - CHU Haut Levêque, Pessac
  - CHU Pontchaillou, Rennes
  - CHU Hautepierre, Strasbourg
  - CHU Toulouse Rangueil, Toulouse
  - CHU Tours, Tours
  - Hôpital Paul Brousse, Villejuif